CLINICAL TRIAL: NCT06623695
Title: Investigation of the Effects of Core Exercises Performed on Stable and Unstable Ground on Selected Skills
Brief Title: Investigation of the Effects of Core Exercises Performed on Stable
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Nurkan Yılmaz, Assoc. Prof. (Sports Scientist), Inonu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IU-SBF-NY-ETK6431-01
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Core Exercises Training
Keywords: core; unstable ground; exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants were divided into three groups: Stable Ground Group (SGG), Unstable Ground Group (USGG) and Control Group (CG). SGG and USGG exercise participants participated in a core exercise program for a total of 25-30 minutes, 2 days a week for 5 weeks. SGG participants performed exercises on a stable floor surface, while USGG participants completed the exercise program on a bosuball. CG did not participate in any exercise program. CG continued their daily routine activities and maintained their current physical activity levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stable Ground Group (SGG) (Experimental): Stable Ground Group (SGG) participants performed exercises on a stable floor surface
  Interventions: Other: Exercise
- Unstable Ground Group (USGG) (Experimental): Unstable Ground Group (USGG) participants completed the exercise program on a bosuball.
  Interventions: Other: Exercise
- Control Group (CG) (No Intervention): Control Group (CG) did not participate in any exercise program. CG continued their daily routine activities and maintained their current physical activity levels.

INTERVENTIONS:
Other: Exercise — SGG performed the exercise program on a fixed ground surface. SGG exercise participants participated in a core exercise program for a total of 25-30 minutes, 2 days a week for 5 weeks.
  Arms: Stable Ground Group (SGG)
Other: Exercise — USGG participants completed the exercise program on a bosuball. USGG exercise participants participated in a core exercise program for a total of 25-30 minutes, 2 days a week for 5 weeks.
  Arms: Unstable Ground Group (USGG)

SUMMARY:
The popularity of core stability and strengthening exercise programs in physical rehabilitation and fitness practice, which has become popular since the 20th century, is increasing day by day. The purpose of this research is to reveal the effects of core stability and core strength exercises performed on stable and unstable ground on selected skills.

DETAILED DESCRIPTION:
Scientific studies have shown that there is no clear view on the effects of core exercise models applied on different surfaces, and there are very few studies that observe performance increases in sports activities. Based on this, the aim of this study is to understand more clearly the effects of core stability and core strength exercises performed on stable and unstable ground on selected skills and to implement more functional training programs accordingly. Thus, it is assumed that core training will provide strong positive effects on performance in both athletic and daily activities.

Methods A total of 31 young individuals aged between 18-23, studying at Malatya Inonu University Faculty of Sports Sciences and without any health problems, were included in the study. Participants were divided into three groups: Stable Ground Group (SGG), Unstable Ground Group (USGG) and Control Group (CG). SGG and USGG exercise participants participated in a core exercise program for a total of 25-30 minutes, 2 days a week for 5 weeks. SGG participants performed exercises on a stable floor surface, while USGG participants completed the exercise program on a bosuball. . CG did not participate in any exercise program. CG continued their daily routine activities and maintained their current physical activity levels. The testers were blind to the group (control or training) each subject allocated to. At the end of the exercise protocol, the same procedures applied for the pre-test were applied for the post-test measurements. All tests were performed in an indoor sports hall. All data obtained were recorded on a form created specifically for the study.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy,
* Having never done core exercise before,
* Being 18 years old or older,
* Being a volunteer

Exclusion Criteria:

* Having any injury,
* Not participating in the core training program regularly in this study,
* Being injured during the training application phase.

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Hand Grip Strength Test | 5 weeks
  For the measurement, Takei A5401/Japan brand digital hand dynamometer was used. This dynamometer is a digital hand dynamometer with an adjustable grip arm that can measure between 5.0 kg/lb -100.0 kg/lb with a precision of 0.1 kg. Before starting the measurements, the dynamometer was adjusted according to the participants' hand sizes and during the measurements, the participants were asked to stand in a standing position, with their feet shoulder-width apart, their elbows in full extension and their arms not touching the body and facing forward at a 45-degree angle in abduction. During the test, participants were asked not to hold their breath and not to shake the dynamometer by holding it tightly, and then they were asked to squeeze the grip handle with all their strength for 3 seconds (sec), saying one, two, three. Measurements for both hands were repeated 3 times with at least 15 seconds between each trial, and the best performance was recorded in kilograms (kg).
Trunk Lateral Flexion | 5 weeks
  Participants were in a standing position with their feet slightly apart and parallel to each other, and their arms close to and next to the body. For both hands, after the point where the distal tip of the 3rd finger (middle) comes to the thigh is marked, the individual performs lateral flexion and the point where the distal tip of the 3rd finger (middle) comes to is marked again. The distance between two specified points was measured and recorded in cm. The measurements were taken three times for both hands, and the highest value was recorded as the result.
Trunk Extansion | 5 weeks
  Participants stood facing the wall, with their pelvis and entire body touching the wall. For the measurement, the participant performed trunk extension by moving his/her head back from the wall without breaking contact with the wall. Thus, the distance between the sternal prominence and the wall was measured with a tape measure and recorded. Then, the participant was supported by supporting the pelvic area and asked to push his/her trunk backwards from the waist area as far as possible. At the last point, the distance between the sternal notch and the wall was measured again. The difference between the first and last values obtained was written on the form in cm. The measurements were made three times and the highest value was recorded as the result.
Sit and Reach | 5 weeks
  Flexibility was measured using a sit-and-reach test, using a sit-and-reach box (Baselıne/ Fabrication Enterprises, Inc., PO Box 1500, White Plains, NewYork). The subjects sat with their feet approximately hip-wide against the testing box (height 30.5 cm.). For the test performance, the subjects was placed seated on the floor with the legs stretched, barefooted and with the soles of the foot attached to the Seat and Reach case. They kept their knees extended and placed the right hand over the left, and slowly reached forward as far as they could by sliding their hands along the measuring board. Participants held this position for approximately 2 sec. and were told that lowering their heads to the lowest point, looking down at the floor, would increase the distance reached. A tape measure on top of the measuring board indicated in centimeters how far beyond the toes each individual reached. The score [in centimeters (cm)]is the greatest distance contacted by the fingertips past the toes
Standing Long Jump Forward Test | 5 weeks
  In the standing long jump test, which is considered a general indicator of muscle condition, participants waited with their feet just behind the starting line before the test began. Then, for the measurement, the participants were instructed to jump as far as possible from the starting line by swinging their arms. They performed 3 trials with 2-minute rest intervals. The distance from the starting line to the farthest point she/he could jump to the landing point at heel contact was measured with a tape measure and the highest distance was recorded in cm.
Bent Arm Hanging | 5 weeks
  The test participants stood in front of a barre apparatus, a platform that could be adjusted according to their height. Participants demonstrated appropriate and comfortable bar grip (prone-supine) style after being informed about the test protocol. During the measurement, the participants were asked to stand on the bar machine for as long as possible with their arms at maximum elbow flexion and their chins hanging above the bar level, and the test was ended when the participants' chins dropped below the bar. The time spent in this position was determined using a stopwatch and recorded as a score in seconds. The test was administered once.
Biering Sorenson Test | 5 weeks
  In the Biering Sorensen test, also known as the trunk extension test, participants were informed about the test protocol. For the measurement, participants were asked to lie face down on the stretcher. Participants were instructed to hang their upper body (hands, arms, head, trunk) down from the stretcher to the level of their anterior superior iliac heads, and lie face down on the stretcher with their lower limbs immobilized (with straps or people). Participants were allowed to place their hands on the chair in front of them before starting the test to avoid getting tired in this position. For the measurement, participants were instructed to remove their hands from the chair, cross their arms in front of their chest, and then lift their upper body until their torso was horizontal to the floor and in line with the stretcher. The time was started when the subject reached the starting position. Participants were instructed to maintain a horizontal body position for as long as possible.
Hexagonal Agility Test | 5 weeks
  A hexagonal shape consisting of six side edges, each side 66 cm long, was drawn on a non-slip surface. Participants were informed about the test protocol. The participant was then asked to move to the center point within the hexagon and take a position facing side A. It was also asked to face point A throughout the test period. The stopwatch starts with the start command and the participant is asked to jump off the line with both feet, starting from line A, over each side line (B, C, D, E, F) and return to the center. The horizontal jumps in and out starting from side A and ending at side A were accepted as 1 round and 3 rounds were performed in this way. If the participant jumps or steps on the wrong line, the test is repeated. At the end of 3 correctly performed laps, the stopwatch was stopped and the elapsed time was recorded. Participants were given two trials after the adaptation phase. The best score was recorded in sec.

CONTACTS AND LOCATIONS:
Overall Officials: Nurkan Yilmaz, Assoc. Prof., Principal Investigator — Inonu University Faculty of Sports Sciences
Locations (1):
- Inonu University Faculty of Sports Sciences Sports Hall, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No